CLINICAL TRIAL: NCT00368862
Title: Phase Four Double-Blind Randomized Comparative Study on Thestudy on the Efficacy of Memantine Hydrochloride and Escitalopram for the Treatment of Co-Morbid Depression and Alcoholism
Brief Title: Efficacy Study of Memantine Hydrochloride and Escitalopram for the Treatment of Co-Morbid Depression and Alcoholism.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Finnish Foundation for Alcohol Studies (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KTL172-9
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2006-08-29 (Estimated); Status verified 2006-08

CONDITIONS: Alcoholism; Depression
Keywords: Alcoholism; Depression; Efficacy study; Memantine; Escitalopram
MeSH Terms: conditions — Alcoholism; Depression | interventions — Memantine; Dexetimide; Escitalopram

INTERVENTIONS:
Drug: Ebixa (memantine hydrochloride)
Drug: Cipralex (escitalopram)

SUMMARY:
The aim of the present study was to examine the influence of memantine, a noncompetitive NMDA receptor blocker, in depression co-morbid with long term alcohol heavy use comparing to SSRI-inhibitor, escitalopram. Second goal is to compare their influence to cognitive tasks and the third goal is to follow up alcohol-use with these two medicines.

DETAILED DESCRIPTION:
Context Depression is common clinical problem among alcoholics and its treatment has no standard and is controversy. Glutamate NMDA-receptors may mediate the effects of long term alcohol related depression and thus the NMDA-receptor modulator memantine could have effects on it.

Objectives The preliminary aim of this study was to identify possible new treatment for depression of alcoholics and compare the efficacy of escitalopram and memantine in co-morbid depression of alcoholism.

Design and setting Double-blind, randomized, naturalistic study, 26-week trial on alcohol dependent outpatients.

Participants Eighty alcohol dependent depressive adults

Intervention Subjects were randomized 1:1 to receive memantine or escitalopram 20 mg per day. During the study the patient received routine psychosocial treatment at A-Clinic. No concomitant intervention on alcohol consumption and no imposed treatment goals. The patients were met weekly in first month, then after 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. The subject/patient is able to read and understand the subject/patient information sheet.
2. Prior to any screening procedures, the subject/patient must have signed the informed consent form. No study-related procedures may be performed before the subject/patient has signed the form.
3. Age 25-70 years
4. Heavy alcohol consumption (males more than 5 doses/ day, female more than 4 doses/day) for at least 10 years
5. Alcohol dependence (DSM-IV) assessed by SCID-I interview.
6. Major depression (DSM-IV) assessed by SCID-I interview. At least 4 weeks past from the previous inpatient treatment for AWS (alcohol withdrawal syndrome).

Exclusion Criteria:

1. Other drug dependence (screened by urine test)
2. Other serious mental illness (DSM-IV)
3. Hazard of suicide
4. Pregnancy
5. Serious kidney, hart or thyroid problem
6. The subject/patient, in the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any reason.
7. Liver cirrhosis or liver enzymes ASAT tai ALAT >200.
8. The person that met the criteria stated in the Finnish Law on Clinical Studies, paragraph 7-10§ (children, pregnant, imamates or mentally handicapped).

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-12; Study Completion 2006-06

PRIMARY OUTCOMES:
Primary outcomes were MADRS (depression), HAM-A (anxiety), CERAD (cognitive test) and alcohol consumption (time line follow backup).

SECONDARY OUTCOMES:
BDI (depression), BAI (anxiety), OCDS (obsessive-compulsive drinking scale), AUDIT (alcohol use disorder identification) , and SOFAS (social and occupational functions) and quality of life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Hannu E Alho, MD, PhD, Study Director — National Public Health Institute, Department of Mental health and Alcohol Research
Locations (1):
- National Public Health Institute, Department of Mental Health and Alcohol Research, Helsinki, POB 33, Finland

REFERENCES:
- [Result] Maler JM, Esselmann H, Wiltfang J, Kunz N, Lewczuk P, Reulbach U, Bleich S, Ruther E, Kornhuber J. Memantine inhibits ethanol-induced NMDA receptor up-regulation in rat hippocampal neurons. Brain Res. 2005 Aug 9;1052(2):156-62. doi: 10.1016/j.brainres.2005.06.017. PMID 16009352
- [Derived] Muhonen LH, Lahti J, Sinclair D, Lonnqvist J, Alho H. Treatment of alcohol dependence in patients with co-morbid major depressive disorder--predictors for the outcomes with memantine and escitalopram medication. Subst Abuse Treat Prev Policy. 2008 Oct 3;3:20. doi: 10.1186/1747-597X-3-20. PMID 18834506
- [Derived] Muhonen LH, Lonnqvist J, Juva K, Alho H. Double-blind, randomized comparison of memantine and escitalopram for the treatment of major depressive disorder comorbid with alcohol dependence. J Clin Psychiatry. 2008 Mar;69(3):392-9. doi: 10.4088/jcp.v69n0308. PMID 18348597